CLINICAL TRIAL: NCT06959940
Title: Alternative Method to Reduce Pain, Anxiety, Fatigue, and Thirst: Chewing Gum in Labor
Brief Title: Alternative Method: Chewing Gum in Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Nilgun Avci, Assistant professor, PhD, Biruni University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chewing gum in labor
Record Dates: First submitted 2023-11-13; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2023-11

CONDITIONS: Labor Pain
Keywords: Labor; gum; pain; anxiety; fatigue; thirst
MeSH Terms: conditions — Labor Pain; Pain; Anxiety Disorders; Fatigue

STUDY DESIGN:
Intervention Model Description: Power analysis was used to determine the sample. The power of the test was calculated with the G*Power 3.1 program. The effect size in the interventional study conducted by Gundogdu (2019) on pregnant women was based on 0.932. In order to exceed the 95% value in determining the power of the study, it was determined that 94 people, including at least 47 people in the groups, should be reached the 5% significance level and 0.95 effect size (df=0.75; t=1.676).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- This research is planned with experimental design (Experimental): After the pregnant woman in the control group was admitted to the delivery room, the data collection tools "Personal Information Form" and "Pregnant Follow-up Form" were applied. Pregnancy Follow-up Form consists of pain, anxiety, fatigue and thirst scales. The VAS pain, anxiety, fatigue, and thirst scales contains numbers evenly spaced (0-10) on a line. It is an evaluation scale filled out by patients stating their current pain, anxiety, fatigue, and thirst level by giving a number. The cut-off point of the VAS anxiety and thirst scales were found to be four. In VAS anxiety, scores above this cut-off point indicate deviation from normal and individuals must be handled by professionals. IN VAS thirst, patients who score above this score are considered to be experiencing dehydration symptoms.
  Interventions: Other: experimental group (gum group)

INTERVENTIONS:
Other: experimental group (gum group) — After the pregnant woman in the experimental group was admitted to the delivery room, the data collection tools "Personal Information Form" and "Pregnant Follow-up Form" were applied. Pregnant women who agreed to participate in the study were given information about chewing gum. Pain, anxiety, fatigue and thirst scales were administered to the pregnant woman before she started chewing gum. The pregnant woman was allowed to chew gum for 15 minutes. At the end of 15 minutes, the measurements were repeated. Applications were repeated as stated above every two hours until the pregnant woman's dilation reached 5 cm. Routine medical treatment of pregnant women continued.

SUMMARY:
This study is a clinical trial. It aimed to examine the effects of chewing gum on pain, anxiety, fatigue, and thirst in pregnant women (47 experiments; 47 controls) in the first stage of labor. Criteria for inclusion in the study: Pregnant women who gave birth vaginally; voluntarily accept to participate in the research. Exclusion criteria from the study: Pregnant women who have auditory or mental health problems; whose baby dies during labor, who with cervical dilatation of 5 cm or more, who receiving epidural anesthesia, do not like chewing gum, have difficulty chewing, such as weak/loose-fitting dentures. The pain, anxiety, fatigue, and thirst levels of the pregnant women in the control group were evaluated with scales every two hours until their dilatation reached 5 cm. Pregnant women in the experimental group chewed gum and their pain, anxiety, fatigue and thirst levels were evaluated with scales every two hours until their dilation reached 5 cm.

The main questions it aims to answer are:

* Chewing gum during labor is not effective in reducing pain, anxiety, fatigue, and thirst levels.
* Chewing gum during labor; It is effective in reducing the level of pain.
* Chewing gum during labor; It is effective in reducing anxiety.
* Chewing gum during labor; It is effective in reducing thirst.
* Chewing gum during labor; It is effective in reducing fatigue. Routine medical treatment of pregnant women continued all groups. Only pregnant women who in the experimental group chewed gum also.

DETAILED DESCRIPTION:
Objective: In this study, it was aimed to examine the effects of chewing gum on pain, anxiety, fatigue and thirst in pregnant women in the first stage of normal labor.

Methods: The study was conducted in a randomized controlled experimental manner. The universe consisted of all pregnant women who applied to the delivery room of a public institution between April and November 2022. Power analysis was used to determine the sample. 94 pregnant women (47 experiments;47 controls) were included in the study. The study was started after the approval of the ethics committee and the institution. As a data collection tool in the research;"Personal Information Form","Gum Chewing Follow-up Form" and "Pregnant Follow-up Form" were used.

ELIGIBILITY:
Inclusion Criteria:

* Vaginal delivery,
* Who volunteered to participate in the research

Exclusion Criteria:

* Have auditory or mental health problems,
* The baby dies during labour,
* Cervical dilatation of 5 cm or more,
* Receiving epidural anaesthesia,
* People who don't like chewing gum,
* Chewing difficulties due to weak/loose prostheses

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
2 | Anxiety scale used starting to chew gum. Then after chewing gum (immediately after the intervention), the scale was repeated. The score on the scale is between 0-10, just like the VAS (visual analogue pain scale). The higher score is the greater problem.
  Change from anxiety scale scores at control group or experimental group in during labor
1 | Pain scale used starting to chew gum. Then after chewing gum (immediately after the intervention), the scale was repeated. The score on the scale is between 0-10, just like the VAS (visual analogue pain scale). The higher score is the greater problem.
  Change from pain scale scores at control group or experimental group in during labor
3 | Fatigue scale used starting to chew gum. Then after chewing gum (immediately after the intervention), the scale was repeated. The score on the scale is between 0-10, just like the VAS (visual analogue pain scale). The higher score is the greater problem.
  Change from fatigue scale scores at control group or experimental group in during labor
4 | Thirst scale used starting to chew gum. Then after chewing gum (immediately after the intervention), the scale was repeated. The score on the scale is between 0-10, just like the VAS (visual analogue pain scale). The higher score is the greater problem.
  Change from thirst scale scores at control group or experimental group in during labor

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF